CLINICAL TRIAL: NCT00891761
Title: A Study of Single Dose Intravenous Casopitant in Combination With Ondansetron and Dexamethasone for the Prevention of Cisplatin-Induced Nausea and Vomiting
Brief Title: A Study of IV Casopitant for the Prevention of Nausea and Vomiting Caused By Cisplatin-Based Highly Emetogenic Chemotherapy
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study has been cancelled prior to enrollment.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 112512
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Cancer; Chemotherapy-Induced Nausea and Vomiting; Nausea and Vomiting; Solid Tumor Cancer
Keywords: cisplatin; nausea; vomiting; cancer; lung cancer
MeSH Terms: conditions — Neoplasms; Vomiting; Nausea; Lung Neoplasms | interventions — Dexamethasone; casopitant; Exercise; Ondansetron

ARMS (2):
- Active Comparator (Active Comparator): Patients receive IV casopitant (active), IV ondansetron and oral dexamethasone on Day 1 as well as oral dexamethasone on Days 2-4 of each cycle of cisplatin-based highly emetogenic chemotherapy for the prevention of chemotherapy induced nausea and vomiting.
  Interventions: Drug: Dexamethasone; Drug: IV casopitant (active); Drug: Ondansetron
- Placebo Comparator (Placebo Comparator): Patients receive IV casopitant (placebo), IV ondansetron and oral dexamethasone on Day 1 as well as oral dexamethasone on Days 2-4 of each cycle of cisplatin-based highly emetogenic chemotherapy for the prevention of chemotherapy induced nausea and vomiting.
  Interventions: Drug: Dexamethasone; Drug: IV casopitant (placebo); Drug: Ondansetron

INTERVENTIONS:
Drug: Dexamethasone — 16 mg administered orally within 75 minutes prior to the initiation of cisplatin on Day 1, followed by 8 mg doses twice daily (bid) at approximately 12+/-4 hour intervals on days 2, 3, and 4, starting at approximately the same time of day as the Day 1 dose was administered.
  Arms: Active Comparator
Drug: Dexamethasone — 20 mg administered orally within 75 minutes prior to the initiation of cisplatin on Day 1, followed by 8 mg doses twice daily (bid) at approximately 12+/-4 hour intervals on days 2, 3, and 4, starting at approximately the same time of day as the Day 1 dose was administered.
  Arms: Placebo Comparator
Drug: IV casopitant (placebo) — IV casopitant (placebo) administered within 75 minutes prior to the start of cisplatin-based highly emetogenic chemotherapy on study day 1.
  Arms: Placebo Comparator
Drug: IV casopitant (active) — Single-dose 90 mg IV casopitant administered within 75 minutes prior to the start of cisplatin-based highly emetogenic chemotherapy on study Day 1.
  Arms: Active Comparator
Drug: Ondansetron — 32mg IV ondansetron administered over not less than 15 minutes, with administration started and completed within the 75 minutes prior to the initiation of cisplatin therapy on study Day 1.

SUMMARY:
This is a phase III study designed to demonstrate the superiority of single-dose 90 mg intravenous (IV) casopitant over placebo, each in combination with ondansetron and dexamethasone, for the prevention of emesis over the first 0-120 hours (overall phase) following initiation of the cisplatin infusion in the first cycle of highly emetogenic chemotherapy (HEC). Eligibility is limited to subjects who are scheduled to receive their first cycle of chemotherapy which includes at least 60 mg/m2 of cisplatin administered on Day 1 only of a 21 day or 28 day cycle. All subjects will receive IV ondansetron and oral dexamethasone on Day 1 prior to initiation of the cisplatin infusion, followed by oral dexamethasone on Days 2-4. Additionally, subjects will be randomized to receive single-dose 90 mg IV casopitant or matching placebo prior to initiation of a cisplatin-based HEC regimen.

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered eligible for initial inclusion in this study, and progression into subsequent cycles of therapy within the study, only if all of the following criteria apply:

* Subject understands the nature and purpose of this study and the study procedures and has signed an informed consent form for this study to indicate this understanding.
* At least 18 years of age.
* Is scheduled to receive oxaliplatin at a dose between 85 mg/m2 and 130 mg/m2 in their first cycle of therapy for the treatment of colorectal cancer, administered as a single IV dose over 2-6 hours on Day 1 only, in combination with 5FU/LV, or in combination with capecitabine. Refer to Section 4.1 for the list of chemotherapy agents that may be added to oxaliplatin.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2.
* Hematologic and metabolic status adequate for receiving an oxaliplatin-based moderately emetogenic regimen and meeting the following criteria:
* Total Neutrophils ≥1500/mm3 (Standard units : ≥1.5 x 109/L)
* Platelets ≥100,000/mm3 (Standard units: ≥100.0 x 109/L)
* Bilirubin ≤1.5 x upper limit of normal (ULN)
* Serum Creatinine ≤1.5 mg/dL (Standard units : ≤132.6 µmol/L) OR
* Creatinine clearance ≥60 mL/min

Creatinine clearance must be calculated using the Cockcroft-Gault formula:

Clcreat (ml/min) = (140-age [yr]) x body wt [kg] / 72 x serum creatinine [mg/dl] For females: multiply creatinine clearance by a factor of 0.85. OR Clcreat (ml/min) = K x (140-age [yr]) x body wt [kg] / serum creatinine [µmol/L] K=1.05 for females K=1.23 for males

* Liver enzymes must be below the following limits:
* Without known liver metastases: Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤2.5 x ULN.
* With known liver metastases: AST and/or ALT ≤5.0 x ULN.
* Is willing and able to complete daily components of the Subject Diary for Cycle 1 and Cycle 2 without assistance from others.
* A female subject is eligible to enter and participate in this study if she is of:
* non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal. For purposes of this study, postmenopausal is defined as one year without menses)
* child-bearing potential: must have a negative serum pregnancy test result or negative urine dipstick pregnancy test within 24 hours prior to the first dose of investigational product on Cycle 1 Day 1. Women of childbearing potential must also commit to consistent and correct use of an acceptable method of birth control. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:
* male partner who is sterile prior to the female subject's entry into the study and is the sole sexual partner for that female subject;
* oral contraceptives (e.g., oral, injectable, or implantable) with double-barrier method of contraception consisting of spermicide with either condom or diaphragm for a period after the trial to account for a potential drug interaction (minimum of six weeks);
* double-barrier method of contraception consisting of spermicide with either condom or diaphragm;
* intra-uterine device with a documented failure rate of less than 1% per year;
* complete abstinence from intercourse for two weeks before exposure to the investigational product throughout the clinical trial, and for a period after the trial to account for elimination of the drug (minimum of 3 days);
* if subject indicates they will remain abstinent during the period described above, they must agree to follow GSK guidelines for the consistent and correct use of an acceptable method of birth control should they become sexually active.

Exclusion Criteria:

A subject will not be eligible for initial inclusion in this study if any of the following criteria apply, or will not be eligible for subsequent cycles of therapy if any of the following criteria become applicable:

* Has received cytotoxic chemotherapy prior to the first study cycle of chemotherapy, with the exception that previous adjuvant therapy with 5FU/LV or capecitabine is permitted, provided that the last dose of adjuvant therapy was completed at least 6 months prior to receiving the first dose of study medication or investigational product. Previous biological or hormonal therapy completed at any time is permitted.
* Scheduled to receive chemotherapy with any cytotoxic agents (e.g., irinotecan, gemcitabine) or biological agents (e.g., cetuximab, panitumimab) other than the protocol allowed chemotherapy described in Inclusion Criterion 3.
* Is a female subject who is pregnant or lactating.
* Has received radiation therapy in the 10 days prior to the first dose of study medication or investigational product and/or is scheduled to receive such radiation therapy in the 6 days following the first dose of study medication or investigational product in the first cycle of chemotherapy. Radiation therapy may be added in subsequent cycles of chemotherapy.
* Has experienced emesis (i.e., vomiting and/or retching) or clinically significant nausea in the 24 hours preceding the first dose of study medication or investigational product for each cycle of chemotherapy.
* Has known central nervous system metastasis, unless previously successfully treated with excision or radiation, and has been stable for at least 1 week immediately prior to receiving the first dose of study medication or investigational product.
* Has increased intracranial pressure, hypercalcemia, an active systemic infection, or any uncontrolled medical condition (other than malignancy) which in the opinion of the Investigator may confound the results of the study, represent another potential etiology for emesis and nausea (other than CINV) or pose an unwarranted risk to the subject.
* Has a known hypersensitivity or contraindication to ondansetron, another 5-HT3 receptor antagonist, dexamethasone, or any component of casopitant.
* Has received an NK-1 receptor antagonist prior to the first study cycle of chemotherapy.
* Has received an investigational drug within the previous 30 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study medication or investigational product, or is scheduled to receive any investigational drug other than casopitant/placebo during the study period.
* Has taken/received any medication of moderate or high emetogenic potential (including antineoplastic agents [see Appendix 2]) within the 48 hours prior to the first dose of study medication or investigational product in each cycle. However, opioid narcotics will be permitted if the subject has been on such medication for at least 7 days at a stable dose prior to the start of each cycle, and has not experienced emesis or nausea from the narcotics.
* Has taken/received any medication with known or potential antiemetic activity within the 24-hour period (unless otherwise stated) prior to receiving the first dose of study medication or investigational product or is expected to require use of such medication during the 120 hour assessment period for Cycle 1 of therapy only. This includes, but is not limited to:
* 5-HT3 receptor antagonists (e.g., additional ondansetron, or granisetron, dolasetron, tropisetron, ramosetron). Palonosetron is not permitted within 7 days prior to administration of study medication or investigational product;
* benzamide / benzamide derivatives (e.g., metoclopramide, alizapride);
* benzodiazepines (except if the subject is receiving such medication for sleep or anxiety and has been on a stable dose for at least 7 days prior to the first dose of investigational product; however, lorazepam is prohibited 24 hours prior to receiving study drug regardless of reason for use);
* phenothiazines (e.g., prochlorperazine, promethazine, fluphenazine, perphenazine, thiethylperazine, chlorpromazine);
* butyrophenones (e.g., haloperidol, droperidol);
* corticosteroids within 72 hours prior to the first dose of study medication or investigational product (e.g., dexamethasone, methylprednisolone); with the exception that topical steroids for skin disorders including eye and ear drops, and inhaled steroids for respiratory disorders at no more than 10 mg prednisone daily or its equivalent are permitted;
* anticholinergics (e.g., scopolamine); with the exception that anticholinergics for the treatment of respiratory disorders and the management of diarrhea (e.g., ipratropium bromide, and hyoscyamine) and anticholinergic eye drops are permitted;
* first-generation antihistamines (e.g., cyclizine, hydroxyzine, diphenhydramine) except for topical use which is permitted;
* domperidone;
* cannabinoids;
* mirtazapine;
* olanzapine.
* Has taken/received strong or moderate inhibitors of CYP3A4 and CYP3A5 for a specified period prior to administration of investigational product in each cycle of therapy.
* Has taken/received inducers of CYP3A4 and CYP3A5 within 14 days prior to the administration of investigational product in each cycle of therapy.
* Is currently taking, or plans to take the following CYP2C8 substrates at any time during the study: the anti-diabetic agent repaglinide or the diuretic torsemide.
* Is currently taking, or plans to take any of the following CYP3A4 substrates at any time during the study: astemizole, cisapride, pimozide, terfenadine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-07 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieve a complete response (defined as no vomiting/retching and no rescue therapy). | Overall phase (0-120 hours) following initiation of the first cycle of a cisplatin-based HEC regimen.

SECONDARY OUTCOMES:
The proportion of subjects who vomit/retch | Acute, delayed and overall phases of Cycle 1
The proportion of subjects who receive anti-emetic rescue medication | Acute, delayed and overall phases of Cycle 1
Maximum nausea score (to assess the severity of nausea), assessed by a Visual Analogue Scale (VAS). | Acute, delayed and overall phases of Cycle 1
The proportion of subjects reporting significant nausea, defined as a maximum nausea score of at least 25 mm on the VAS. | Acute, delayed and overall phases of Cycle 1
The proportion of subjects who achieve a complete response | Acute (0-24 hrs) and delayed (24-120 hrs) phases of Cycle 1
The proportion of subjects reporting nausea, defined as a maximum nausea score of at least 5 mm on the VAS. | Acute, delayed and overall phases of Cycle 1
The proportion of subjects achieving complete protection, defined as complete responders who had no significant nausea. | Acute, delayed and overall phases of Cycle 1
The proportion of subjects achieving total control, defined as complete responders who had no nausea. | Acute, delayed and overall phases of Cycle 1
Time to first anti-emetic rescue medication. | Acute, delayed and overall phases of Cycle 1
Time to first emetic event. | Acute, delayed and overall phases of Cycle 1
Time to loss of complete response. | Acute, delayed and overall phases of Cycle 1
The proportion of subjects who achieve a complete response. | Extended overall phase (0-216 hrs) of Cycle 1
The proportion of subjects who achieve a complete response. | Overall (0-120 hrs), acute and delayed phases of Cycle 2
The impact on subjects' daily life activities, as assessed by the FLIE questionnaire. | Overall phase (0-120 hrs) of Cycle 1.
Assessment of the safety and tolerability of casopitant through routine physical exam, routine clinical laboratory tests, clinical monitoring and AE reporting. | All cycles

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (2):
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Robbinsdale, Minnesota
- GSK Investigational Site, Sherbrooke, Quebec, Canada